CLINICAL TRIAL: NCT00470002
Title: Effects of Growth Hormone (GH) on Parameters of the Nitric Oxide (NO) Pathway
Brief Title: Effects of Growth Hormone on the Nitric Oxide Pathway
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Pharmacia (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MES 03069; VP2-3900-4021576; IRB#3444
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Cardiovascular Disease
Keywords: growth hormone; nitric oxide; nitrate; cyclic guanosine monophosphate; insulin-like growth factor-1; asymmetric dimethylarginine; blood pressure; endothelial progenitor cells
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Somatropin

SUMMARY:
The purpose of the study is to determine whether the treatment with growth hormone has an influence on the nitric oxide pathway in healthy males.

DETAILED DESCRIPTION:
Nitric oxide (NO) is a potent endogenous vasodilator and has shown to inhibit key processes of atherosclerosis like monocyte adhesion, platelet aggregation, and vascular smooth muscle cell proliferation. Impaired endothelial NO production is a main feature of endothelial dysfunction, which by itself is an early step in the course of atherosclerotic vascular disease.

Recent studies could confirm this close association between parameters of the NO pathway and cardiovascular disease and could further enhance the knowledge on the pathophysiological mechanisms. There is a significant relationship between insulin resistance and the endogenous NO synthase inhibitor asymmetric dimethylarginine (ADMA). Moreover, evidence could be provided that plasma levels of ADMA are a strong and independent predictor of mortality and cardiovascular outcome in haemodialysis patients.

Patients with growth hormone deficiency are characterized by a 1.9 fold higher risk of death from cardiovascular disease. Again, there is good evidence, that alterations of the NO-pathway are involved in this increase of cardiovascular risk. A reduced endogenous systemic production of NO was found in patients with growth hormone deficiency, treatment with recombinant growth hormone normalized NO production. The effects of growth hormone on NO are possibly mediated by insulin-like growth factor-I (IGF-I), which stimulates NO synthesis in vitro. The onset of IGF-I increase in healthy volunteers treated with GH is evident after 12 h, the maximum effect takes place between 5 to 8 days. Also in adults with growth hormone deficiency, the major effects of growth hormone treatment on IGF-I levels are observed within 2 weeks. After discontinuation of growth hormone therapy, IGF-1 levels return to base line within 2-3 days.

The aim of the present study is to further elucidate the in vivo effects of GH on the NO pathway and NO mediated cardiovascular functions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects without recent severe diseases
* Age 50 yrs or older
* Body mass index at or below 30 kg/m2
* Insulin-like growth factor-1 level below 200 ng/ml
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial
* Subjects that are willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* History of any severe hepatic, renal, cardiac, endocrine, metabolic, or malignant diseases
* Requirement for medical drug treatment
* Growth hormone treatment during the last 12 months
* Drug dependence, alcohol or nicotine abuse
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-05; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Urinary nitrate excretion | 10 days

SECONDARY OUTCOMES:
Insulin-like growth factor-1 in serum | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Dirk O Stichtenoth, MD, Study Director — Institute of Clinical Pharmacology, Hannover Medical School
Locations (1):
- Institute of Clinical Pharmacology, Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Boger RH, Skamira C, Bode-Boger SM, Brabant G, von zur Muhlen A, Frolich JC. Nitric oxide may mediate the hemodynamic effects of recombinant growth hormone in patients with acquired growth hormone deficiency. A double-blind, placebo-controlled study. J Clin Invest. 1996 Dec 15;98(12):2706-13. doi: 10.1172/JCI119095. PMID 8981915
- [Background] Tsukahara H, Gordienko DV, Tonshoff B, Gelato MC, Goligorsky MS. Direct demonstration of insulin-like growth factor-I-induced nitric oxide production by endothelial cells. Kidney Int. 1994 Feb;45(2):598-604. doi: 10.1038/ki.1994.78. PMID 7513035